CLINICAL TRIAL: NCT00040014
Title: Open Label, Multicenter, Randomized, Controlled Study of IM or Oral Exemestane (Aromasin) in Postmenopausal Women With Advanced Breast Cancer Having Progressed on Tamoxifen.
Brief Title: Open Label, Multicenter, Randomized, Controlled Study of IM or Oral Exemestane (Aromasin) in Postmenopausal Women
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 971-ONC-0401-003
Record Dates: First submitted 2002-06-18; First posted 2002-06-20 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

INTERVENTIONS:
Drug: exemestane

SUMMARY:
The purpose of this study is to find out if the two different formulations of exemestane (Aromasin), oral and injectable, are equivalent in terms of pharmacodynamics and pharmacokinetics, i.e., if ultimately both formulations have the same efficacy in postmenopausal women with metastatic breast cancer who have failed previous antiestrogens therapy and are equally safe.

ELIGIBILITY:
Inclusion Criteria:

* other diagnosed with breast cancer
* estrogen receptor positivity
* Postmenopausal status
* advanced disease
* progression to previous tamoxifen therapy

Exclusion Criteria:

* more than 1 chemotherapy and / or more than 1 hormonotherapy for advanced disease
* previous hormonotherapy other than Tamoxifen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To determine the pharmacodynamic equivalence at steady state of the IM formulation of exemestane with the oral formulation in terms of plasma estrone sulphate inhibitory effect in postmenopausal women with advanced breast cancer.

SECONDARY OUTCOMES:
to characterize the pharmacodynamic profile of the two formulations in terms of estrogens, androgens, and sec hormone binding globulin
to characterize the pharmacokinetics of exemestane and 17 hydroexemestane after administration of the two formulations
to evaluate the relationships between pharmacokinetics and pharmacodynamics after intramuscular and oral administration of exemestane
to evaluate the efficacy (as tumor response)
to evaluate the incidence and severity of systemic toxicities and of the local tolerability of the injectable formulation
to evaluate the effect on serum bone turnover markers

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Leicester, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=971-ONC-0401-003&StudyName=Open+Label%2C+Multicenter%2C+Randomized%2C+Controlled+Study+of+IM+or+Oral+Exemestane+%28Aromasin%29+in+Postmenopausal+Women